CLINICAL TRIAL: NCT05464433
Title: Open-Label, PhaseIb/Ⅱ Study of Tislelizumab and Mitoxantrone Hydrochloride Liposome Combination Treatment in Patients with Relapsed or Refractory Extranodal Natural Killer/T Cell Lymphoma（ALLIANCE-022）
Brief Title: Tislelizumab Combined with Mitoxantrone Hydrochloride Liposome in Extranodal Natural Killer/T Cell Lymphoma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Qingqing Cai, Chief physician, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2022-300
Record Dates: First submitted 2022-07-04; First posted 2022-07-19 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Extranodal Natural Killer T Cell Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- liposomal mitoxantrone hydrochloride (Experimental): Patients with recurrent and refractory Extranodal Natural Killer/T Cell Lymphoma（NKTCL）will receive sequentially higher doses of liposomal mitoxantrone hydrochloride in combination with tislelizumab for 6 cycles (planned) (28 days per cycle). The initial dose of liposomal mitoxantrone hydrochloride is 16 mg/m2.
  Interventions: Drug: Tislelizumab combined with Liposomal mitoxantrone hydrochloride; Drug: Maintenance of tislelizumab

INTERVENTIONS:
Drug: Tislelizumab combined with Liposomal mitoxantrone hydrochloride — Drug: liposomal mitoxantrone hydrochloride, tislelizumab Drug: Liposomal mitoxantrone hydrochloride (16 mg/m2, 20 mg/m2) will be administered by an intravenous infusion on day 1 of each 28-day cycle.
  Drug: tislelizumab(200 mg) will be taken orally on day 1 of each 28-day cycle.
Drug: Maintenance of tislelizumab — Drug: tislelizumab(200 mg) will be taken orally on day 1 of each 21-day cycle

SUMMARY:
This is a prospective, open-label, single arm, multicenter clinical study to evaluate the safety, tolerability, efficacy in combination with tislelizumab and mitoxantrone hydrochloride liposome combination treatment in patients with relapsed or refractory Extranodal Natural Killer/T Cell Lymphoma（NKTCL）

DETAILED DESCRIPTION:
This is a prospective, open-label, single arm, multicenter clinical study to explore the maximum tolerated dose (MTD) of liposomal mitoxantrone hydrochloride when combined with tislelizumab in patients with relapsed or refractory Extranodal Natural Killer/T Cell Lymphoma（NKTCL）. Liposomal mitoxantrone hydrochloride will be given on day 1 at two different doses (16 mg/m2, 20 mg/m2) and be combined with tislelizumab. The dose limited toxicity (DLT) will be evaluated after the first cycle of therapy. A maximum of 6 cycles of therapy are planned. An dose expansion study of mitoxanquinone hydrochloride liposome at recommended phaseII dose (RP2D) dose level combined with tirelizumab was conducted to explore the efficacy and safety tolerance of the combined regimen. After 6 cycles of induction therapy, if the outcome was assessed as complete remission (CR)/partial remission (PR)/Stable disease (SD), continued maintenance therapy with tirelizumab.

ELIGIBILITY:
Inclusion Criteria:

* 1. Histologically confirmed diagnosis of Extranodal Natural Killer/T Cell Lymphoma（NKTCL）
* 2. Subjects fully understand and voluntarily participate in this study and sign informed consent
* 3. Age ≥18, ≤75 years, no gender limitation
* 4. Relapsed or refractory NKTCL that has failed to be treated with a asparaginase-based chemotherapy or chemoradiotherapy regimen. Refractory definition: I) the efficacy of chemotherapy with asparaginase-containing regimen did not reach CR; Or II) disease progression within 6 months of the last regimen containing asparaginase; Definition of recurrence: lymphoma that recurred after a complete response (CR) was achieved with initial chemotherapy
* 5. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0-2；
* 6. Expected survival ≥ 3 months;
* 7. There must be at least one measurable or evaluable lesion that meets the evaluation criteria for Lugano 2014 lymphoma: measurable lesion: Positron emission tomography / computed tomography (PET/CT) or CT and/or MRI, intranode lesions with long diameter >1.5cm, short diameter >1.0cm, or exnode lesions with long diameter > 1.0 cm; PET CT examination of the lesion showing increased uptake in lymph nodes or extranodal areas (higher than liver) and imaging features consistent with lymphoma can be evaluated.
* 8. Without hemophagocytic syndrome; If patients diagnosed hemophagocytic syndrome are treated with anti-hemophagocytic syndrome drugs, the general physical condition of the patients will be evaluated by the investigator to determine whether the patients can be included in the group.
* 9. The following required baseline laboratory data:

  1. White blood cell，WBC≥3.0×109/L(Bone marrow invasive patient≥2.0×109/L),Absolute neutrophil count，ANC ≥1.5×109/L, （Bone marrow invasive patient≥1.0×109/L) Platelet count (PLT) ≥75×109/L, （Bone marrow invasive patient≥50×109/L) ，Hemoglobin (HB)≥ 80g/L, No granulocyte growth factor, platelet, or red blood cell transfusions were received within 14 days prior to examination.
  2. Total bilirubin (TBIL) ≤1.5×upper limit of normal (ULN) （The liver invasion≤3.0×ULN）Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN , Serum creatinine ，Scr ≤1.5×ULN（The liver invasion≤5.0×ULN）
  3. Renal function：creatinine, Cr≤1.5×ULN
  4. Coagulation function： International Normalized Ratio，INR≤1.5 ×ULN； Prothrombin Time (PT)、Activated Partial Thromboplastin Time (APTT)≤1.5×ULN（Unless the patient is receiving anticoagulant therapy and PT and APTT are within the expected range of anticoagulant therapy at screening time）；
  5. Thyroid stimulating hormone (TSH) or free thyroid hormone (FT4) or free triiodothyronine (FT3) were within 10% of normal value (note: abnormal TSH caused by non-autoimmune causes can be included in the group);

Exclusion Criteria:

* 1. The subject had previously received mitoxantrone liposomes or the total cumulative dose of mitoxantrone is more than 160 mg/m2 and the total cumulative dose of doxorubicin is more than 360 mg/m2
* 2. A history of other malignant tumors within the past 5 years; Or other tumors (except basal cell carcinoma of the skin)
* 3. Invasive NK cell leukemia; Or central nervous system invasion;
* 4. Participated in clinical trials of other drugs within 4 weeks prior to study commencement;
* 5. Patients had received antitumor therapy 4 weeks prior to study initiation;
* 6. Patients who received allogeneic hematopoietic stem cell transplantation within 3 years prior to study drug administration (patients who received allogeneic hematopoietic stem cell transplantation more than 3 years prior to study drug administration and who do not currently have graft-versus-host reaction can be included); Received autologous hematopoietic stem cell 8 transplantation within 100 days prior to administration of the study drug;
* 7. People with a history of Human Immunodeficiency Virus infection and acquired Immunodeficiency syndrome;
* 8. Patients with chronic active hepatitis B or active hepatitis C. Background Hepatitis B Surface Antigen (HBsAg) or Hepatitis B core Antibody (HBcAb) or Hepatitis C Virus (HCV) antibody, Must be further tested for Hepatitis B Virus (HBV) DNA (no more than 1000 copies /mL or 2 00 IU/mL) and HCV RNA (no more than the lower limit of the assay). Active hepatitis B or C infection requiring treatment should be excluded. Hepatitis B virus carriers, stable hepatitis B after drug treatment (DNA should not be more than 1000 copies /mL or 200 IU/mL and cured hepatitis C patients can be included;
* 9. Subjects who required systemic glucocorticoid therapy or other immunosuppressant therapy for a condition within 14 days prior to initiation of treatment [subjects were allowed to use topical, ocular, intra-articular, intranasal, and inhaled glucocorticoid therapy (with very low systemic absorption); It is permissible to use glucocorticoids for short-term (≤ 7 days) prophylactic treatment (e.g., contrast agent allergy) or for the treatment of non-autoimmune diseases (e.g., delayed hypersensitivity from contact allergens)
* 10. With activity, and over the past two years, need systemic treatment of autoimmune diseases (hormone replacement therapy is not considered a systemic treatment, such as type 1 diabetes, by accepting thyroid hormone replacement therapy for hypothyroidism, only need to accept the physiological doses of sugar cortical hormone replacement therapy adrenocortical function is low or pituitary function in patients with low); Patients with autoimmune diseases who have not required systemic treatment within the past two years can be enrolled;
* 11. Heart function and disease meet one of the following conditions:

  1. Long QTc syndrome or QTc interval > 480 MS;
  2. Complete left bundle branch block, grade II or III atrioventricular block;
  3. Serious and uncontrolled arrhythmias requiring drug treatment;
  4. New York Heart Association grade ≥ III;
  5. Cardiac ejection fraction (LVEF)< 50%;
  6. A history of myocardial infarction, unstable angina pectoris, severe unstable ventricular arrhythmia or any other arrhythmia requiring treatment, a history of clinically serious pericardial disease, or ECG evidence of acute ischemia or active conduction system abnormalities within 6 months before recruitment.、
* 12. Patients who underwent major surgery within 28 days before enrollment; Chronic unhealed wounds or broken bones;
* 13. Live attenuated vaccines (excluding influenza vaccines) received within 4 weeks prior to enrollment or planned during the study period;
* 14. Pregnant and lactating women and subjects of childbearing age who do not want to use contraception;
* 15. Mentally ill persons or persons unable to obtain informed consent;
* 16. Active infection, except for tumor-associated symptom B fever.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2022-06-23 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Dose limited toxicities (DLTs) | Cycle 1 (28 days)
  To identify the DLT
Recommended Phase II Dose（RP2D） | Cycle 1 (28 days)
  To identify the RP2D
Complete response rate (CR) | Up to 24 weeks
  To investigate the preliminary antitumor efficacy

SECONDARY OUTCOMES:
Number of participants with adverse events (AE) and severe adverse events (SAE) as assessed by CTCAE v5.0 | Up to 24 weeks
  To identify the incidence of AE and SAE
Overall response rate (ORR) | Up to 24 weeks
  To investigate the preliminary antitumor efficacy
Disease control rate（DCR） | Up to 24 weeks
  To investigate the preliminary antitumor efficacy
Progression-free survival（PFS） | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  To investigate the preliminary antitumor efficacy

OTHER OUTCOMES:
Combined positive score (CPS) as assessed by immunohistochemical (IHC) staining for PD-L1 | Through study completion, an average of 1 year
  To explore the correlation between CPS and response to immunotherapy
Tumor proportion scoring (TPS) as assessed by immunohistochemical (IHC) staining for PD-L1 | Through study completion, an average of 1 year
  To explore the correlation between TPS and response to immunotherapy
Tumor mutation burden (TMB) as assessed by high throughput sequencing | Through study completion, an average of 1 year
  To measure the number of mutations carried by tumor cells and evaluate the correlation between TMB and response to immunotherapy

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Beijing Tongren Hospital, Capital Medical University, Beijing
  - Peking Union Medical College Hospital, Beijing
  - The Second Hospital of Dalian Medical University, Dalian
  - Sun Yat-Sen University Cancer Center, Guangzhou
  - The First Affiliated Hospital/School of Clinical Medicine of Guangdong Pharmaceutical University, Guangzhou
  - Jiangxi Cancer Hospital, Nanchang